CLINICAL TRIAL: NCT00853827
Title: A 104 Week, Randomized, Double Blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy of Aliskiren on the Progression of Atherosclerosis in Patients With Coronary Artery Disease When Added to Optimal Background Therapy
Brief Title: Safety and Efficacy of Aliskiren on the Progression of Atherosclerosis in Coronary Artery Disease Patients
Acronym: AQUARIUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2366; 2008-006447-40
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease (CAD); Coronary Atherosclerosis
Keywords: CAD; coronary artery disease; coronary atherosclerosis; coronary angiography; IVUS; intravascular ultrasound; plasma renin activity; renin angiotensin aldosterone system,; direct renin inhibitors; coronary atheroma
MeSH Terms: conditions — Coronary Artery Disease | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): Aliskiren 300 mg
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: Aliskiren — 300 mg
  Arms: 2

SUMMARY:
The study will assess the change in coronary atherosclerotic disease as determined by intravascular ultrasound (IVUS) for aliskiren compared to placebo when given in addition to standard therapy in patients with coronary artery disease (CAD) and a blood pressure in the pre-hypertensive range.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CAD who have blood pressure in the pre-hypertensive range defined as a msSBP ≥ 125 and ≤ 139mmHg and a msDBP < 90mmHg.
* Patients with or without current treatment for hypertension
* Angiographic evidence of coronary artery disease
* At least 2 qualifying Cardiovascular risk factors at Visit 1

Exclusion Criteria:

* Baseline IVUS determined unacceptable
* Patients requiring treatment with disallowed study medications
* Patients with clinically significant heart disease
* Previous or current diagnosis of heart failure (NYHA Class IV) or a documented left ventricular ejection fraction of < 25%
* Patients requiring treatment with any 2 of the following classes of medication at Visit 1 or Visit 2:

  * Angiotensin converting enzyme inhibitors
  * Angiotensin receptor blockers
  * aldosterone receptor blockers or a direct renin inhibitor.
* Other conditions may apply

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2009-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Director — Novartis
Locations (116):
- United States (51):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Farmington, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Hudson, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Safety Harbor, Florida
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Elkhart, Indiana
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Midland, Michigan
  - Novartis Investigative Site, Petoskey, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Williamsville, New York
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Bend, Oregon
  - Novartis Investigative Site, Hillsboro, Oregon
  - Novartis Investigative Site, Danville, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Oak Ridge, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Katy, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Argentina (4):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Australia (5):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
- Belgium (7):
  - Novartis Investigative Site, Aalst, Belgium
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Anderlecht
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ottignies
- Canada (7):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- France (4):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Plessis-Robinson
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Germany (8):
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuss
- Hungary (5):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Budapest, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Italy (10):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Sesto San Giovanni, MI
  - Novartis Investigative Site, Massa, MS
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Novara
- Poland (4):
  - Novartis Investigative Site, Krakow, Poland
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Warsaw
- Spain (11):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Galdakano, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadanonda, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias

REFERENCES:
- [Derived] Puri R, Nissen SE, Menon V, Shao M, Hsu A, Bakris GL, Kastelein JJ, Williams B, Armbrecht J, Brunel P, Kataoka Y, Nicholls SJ. Effects of aliskiren in diabetic and non-diabetic patients with coronary artery disease: Insights from AQUARIUS. Atherosclerosis. 2015 Dec;243(2):553-9. doi: 10.1016/j.atherosclerosis.2015.10.019. Epub 2015 Oct 20. PMID 26523993
- [Derived] Nicholls SJ, Bakris GL, Kastelein JJ, Menon V, Williams B, Armbrecht J, Brunel P, Nicolaides M, Hsu A, Hu B, Fang H, Puri R, Uno K, Kataoka Y, Bash D, Nissen SE. Effect of aliskiren on progression of coronary disease in patients with prehypertension: the AQUARIUS randomized clinical trial. JAMA. 2013 Sep 18;310(11):1135-44. doi: 10.1001/jama.2013.277169. PMID 23999933

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren: Period 1(Screening Period) visit 1(Day -42 to Day -1) eligibility for study participation was assessed. Period 2: Visit 2 to 3, single blind for 1 week: patients received aliskiren 150 mg. Period 3: visit 3 to 15, Double-blind Randomization/Forced Titration and Maintenance Period for 103 weeks: patients received 2 tablets aliskiren 150 mg (force titration)
- Placebo: Period 1(Screening Period) visit 1(Day -42 to Day -1) eligibility for study participation was assessed. Period 2: visit 2 to 3, single blind for 1 week: patients received 1 tablet aliskiren 150 mg, 1 tablet placebo 150 mg. Period 3: visit 3 to 15, Double-blind Randomization/Forced Titration and Maintenance Period for 103 weeks: patients received 2 tablets placebo 150 mg
Period: Single Blind Period (1 Week)
Arm/Group | Aliskiren | Placebo
Started | 652 (Enrolled patients in single blind) | 0 (This arm was only used in double blind period)
Completed | 613 (Completed patients in single blind period) | 0
Not Completed | 39 | 0
Not completed — Other | 4 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Abnormal laboratory value | 3 | 0
Not completed — Abnormal test procedure result | 1 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 12 | 0
Period: Double Blind Period (103 Weeks)
Arm/Group | Aliskiren | Placebo
Started | 305 ("Started" indicates number of patients in randomized set, full analysis set (FAS) and safety set.) | 308
Modified Full Analysis Set (mFAS) | 225 | 233
Completed | 201 | 199
Not Completed | 104 | 109
Not completed — Adverse Event | 25 | 14
Not completed — Abnormal laboratory values | 0 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Patient's no longer requires study drug | 3 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 19 | 18
Not completed — Lost to Follow-up | 8 | 10
Not completed — Administrative problems | 45 | 56
Not completed — Death | 1 | 6

BASELINE CHARACTERISTICS:
Population: Randomized - All patients who received a randomization number, regardless of whether or not the patient received the trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 305 | 308 | 613
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.35) | 59.2 (8.32) | 59.7 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 69 | 146
  Male | 228 | 239 | 467

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Atheroma Volume(PAV) After 104 Weeks of Treatment
Description: Change from baseline in PAV for all matched slices of anatomically comparable segments of the target coronary artery were assessed by intravascular ultrasound (IVUS) evaluation after 104 weeks of treatment . calculation for change is the value at the later time point minus the value at the earlier time point, with positive numbers to represent increases and negative numbers to represent decreases
Time Frame: Baseline, 104 weeks
Population: Full Analysis Set (FAS) - All randomized patients. Patients were analyzed according to the treatment that they were assigned at randomization. All patients who had a valid baseline and post baseline IVUS measurement and post-baseline IVUS measurement and at least ≥72 weeks of treatment were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of baseline
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 225 | 233
percentage of baseline | -0.33 (0.18) | 0.11 (0.18)

2. Secondary Outcome: Change in Normalized Total Atheroma Volume (TAV) as Assessed by IVUS
Description: Change from baseline in normalized total atheroma volume (TAV) (mm^3) for all matched slices of anatomically comparable segments of the target coronary artery were assess by IVUS after 104 weeks of treatment. calculation for change is the value at the later time point minus the value at the earlier time point, with positive numbers to represent increases and negative numbers to represent decreases
Time Frame: Baseline, 104 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 225 | 233
mm^3 | -4.11 (1.10) | -2.07 (1.09)

3. Secondary Outcome: Patients That Demonstrated Evidence of Atheroma Regression
Description: Atheroma regression is defined as change from baseline to endpoint in PAV <0 .
Time Frame: Baseline to endpoint (104 weeks)
Population: Full Analysis Set (FAS) - All randomized patients. Patients were analyzed according to the treatment that they were assigned at randomization
Measure: Number; unit: Participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 225 | 233
Participants | 128 | 114

4. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events, and Death
Description: overall safety and tolerability of aliskiren 300 mg compared to placebo in patients with CAD and BP in the pre-hypertensive (high normal) range with or without treatment for hypertension following 104 weeks of treatment. Any Adverse Event was defined as occurrence of any symptom regardless of intensity grade, Serious Adverse Event (SAEs) assessed as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in persistent or significant disability/incapacity.
Time Frame: 104 weeks
Population: Safety - All patients who received at least one dose of double-blind trial medication. Patients were analyzed according to the treatment that they received
Measure: Number; unit: Number of patients
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 305 | 308
Number of patients
  SAEs | 76 | 97
  AE | 228 | 227
  Death | 1 | 6

ADVERSE EVENTS:
Groups:
- Aliskiren 300 mg: Visit 2 to 3, single blind for 1 week: patients received aliskiren 150 mg. visit 3 to 15, Double-blind Randomization/Forced Titration and Maintenance Period for 103 weeks: patients received 2 tablets aliskiren 150 mg (force titration)
Arm/Group | Aliskiren 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 76/305 | 97/308
Other Adverse Events (participants affected / at risk) | 186/305 | 175/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=305) | Placebo (N=308)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 6 | 12
Angina unstable (Cardiac disorders) | 6 | 6
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 5
Coronary artery occlusion (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 2 | 5
Myocardial infarction (Cardiac disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 4
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Sweat gland infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 2 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 4
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 2
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral microangiopathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Reperfusion injury (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (N=305) | Placebo (N=308)
Angina pectoris (Cardiac disorders) | 21 | 24
Palpitations (Cardiac disorders) | 4 | 8
Constipation (Gastrointestinal disorders) | 8 | 10
Diarrhoea (Gastrointestinal disorders) | 20 | 15
Dyspepsia (Gastrointestinal disorders) | 5 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 15 | 13
Asthenia (General disorders) | 7 | 8
Chest pain (General disorders) | 5 | 9
Fatigue (General disorders) | 32 | 21
Non-cardiac chest pain (General disorders) | 23 | 21
Oedema peripheral (General disorders) | 19 | 18
Bronchitis (Infections and infestations) | 10 | 14
Influenza (Infections and infestations) | 16 | 10
Nasopharyngitis (Infections and infestations) | 23 | 13
Sinusitis (Infections and infestations) | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Urinary tract infection (Infections and infestations) | 8 | 10
Fall (Injury, poisoning and procedural complications) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 15
Dizziness (Nervous system disorders) | 35 | 28
Headache (Nervous system disorders) | 18 | 22
Hypoaesthesia (Nervous system disorders) | 9 | 7
Syncope (Nervous system disorders) | 9 | 4
Anxiety (Psychiatric disorders) | 3 | 9
Depression (Psychiatric disorders) | 6 | 12
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Hypertension (Vascular disorders) | 16 | 22
Hypotension (Vascular disorders) | 21 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety